CLINICAL TRIAL: NCT00645853
Title: Long-term Treatment With the Oral Direct Thrombin Inhibitor AZD0837, Compared to Vitamin-K Antagonists, as Stroke Prevention in Patients With Non-valvular Atrial Fibrillation and One or More Risk Factors for Stroke and Systemic Embolic Events. A 5-year Follow-up Study
Brief Title: Long-term Safety in Atrial Fibrillation Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D1250C00042
Record Dates: First submitted 2008-03-19; First posted 2008-03-28 (Estimated); Results first posted 2012-03-06 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Persistent or Permanent Nonvalvular Atrial Fibrillation
MeSH Terms: interventions — AZD 0837; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD0837
- 2 (Active Comparator)
  Interventions: Drug: VKA INR 2-3

INTERVENTIONS:
Drug: AZD0837 — Treatment with AZD0837 starting with 4 different doses, 150 mg od, 300 mg od, 200 mg bid or 450 mg od and then switching to one general common dose, 300 mg od
  Arms: 1
Drug: VKA INR 2-3 — Vitamin K antagonists (VKA), titrated to an international normalised ratio (INR) of 2.0 to 3.0 with a target value of 2.5
  Other Names: warfarin
  Arms: 2

SUMMARY:
The purpose of this study is to provide safety and tolerability data for AZD0837 during long-term treatment (5 years) in patients with non-valvular atrial fibrillation (AF) and one or more additional risk factors for stroke and systemic embolic events (moderate to high risk patients).

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal, persistent or permanent Non Valvular Atrial Fibrillation with one or more additional risk factors for stroke and systemic embolic event
* completing treatment with study drug in D1250C00008.

Exclusion Criteria:

* Atrial Fibrillation secondary to reversible disorders, eg hyperthyroidism
* Presence of a valvular heart disease, mechanical heart valves, active endocarditis, left ventricular aneurysm or thrombus, atrial myxoma or any condition other than Atrial Fibrillation requiring chronic anticoagulation treatment
* Myocardial infarction, heart surgery or percutaneous coronary intervention (PCI) within the previous three months prior to inclusion; Stroke and/or systemic embolism within the previous 30 days prior to inclusion
* Conditions associated with increased risk of major bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2007-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Hvilstedt Rasmussen, MD, PhD, FESC, Principal Investigator — Head of Cardiology at Heart Centre Aalborg Aarhus University Hospital DK 9100 Aalborg Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population included male and female participants >18 years of age with chronic non-valvular Atrial Fibrillation. The participants were recruited during the time period from 25 October 2007 to 20 May 2008 at medical clinics in Europe.
Pre-assignment Details: All participants had previously participated in the Prevention of Stroke and Systemic Embolic Events in Patients With Atrial Fibrillation (NCT00684307) study
Groups:
- AZD0837: Treatment with AZD0837 starting with 4 different doses, 150 mg od, 300 mg od, 200 mg bid or 450 mg od, then switching to one general common dose, 300 mg od.
- VKA, INR 2-3: Vitamin K antagonists (VKA), titrated to an international normalised ratio (INR) of 2.0 to 3.0 with a target value of 2.5
Period: Overall Study
Arm/Group | AZD0837 | VKA, INR 2-3
Started | 288 | 235
No of Patients After Dose Switch | 209 (All patients in the AZD0837 arm switched from their initial doses, to a general dose of 300 mg od) | 188 (No changes for VKA patients)
Discontinued Patient No Due to Closure | 196 (No of patients discontinued due the study termination caused tablet formulation stability problems) | 178 (No of patients discontinued due the study termination caused tablet formulation stability problems)
AZ Study Closure in Hungary | 60 | 40
Completed | 196 | 178
Not Completed | 92 | 57
Not completed — Adverse Event | 18 | 7
Not completed — AZ study closure in Hungary | 60 | 40
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Discontinuation criteria | 2 | 2
Not completed — recall of ICF, planned operation, death | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD0837 | VKA, INR 2-3 | Total
Number analyzed (Participants) | 288 | 235 | 523
Age Continuous [Mean (Full Range); unit: Years] | 69.9 [34 to 93] | 68.0 [33 to 86] | 68.95 [33 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 73 | 163
  Male | 198 | 162 | 360

OUTCOME MEASURES:

1. Primary Outcome: Bleeding: Number of Patients With Any Bleeding Event, During Treatment Period
Description: Participants
Time Frame: 154-711 days on treatment
Measure: Number; unit: Participants
Arm/Group | AZD0837 | VKA, INR 2-3
Number analyzed (Participants) | 288 | 235
Participants | 55 | 56

2. Secondary Outcome: Alanine Transaminase (ALAT): Number of Patients With ALAT>=3xULN, Post Baseline
Description: ULN=Upper limit of Normal
Time Frame: From baseline to Follow up
Measure: Number; unit: Participants
Arm/Group | AZD0837 | VKA, INR 2-3
Number analyzed (Participants) | 288 | 235
Participants | 9 | 6

3. Secondary Outcome: Bilirubin: Number of Patients With Bilirubin>=2xULN, Post Baseline
Time Frame: From baseline to Follow up
Measure: Number; unit: Participants
Arm/Group | AZD0837 | VKA, INR 2-3
Number analyzed (Participants) | 288 | 235
Participants | 3 | 3

4. Secondary Outcome: Creatinine: Absolute Change From Baseline, at End of Treatment
Time Frame: Baseline and End of treatment
Measure: Mean (Full Range); unit: µmol/L
Arm/Group | AZD0837 | VKA, INR 2-3
Number analyzed (Participants) | 288 | 235
µmol/L | 3.70 (-67.0) [-67.0 to 120.0] | -1.17 (-56.0) [-56.0 to 116]

5. Secondary Outcome: D-dimer:Median and Quartile Range at End of Treatment
Description: Median (Lower Quartile-Upper Quartile ), ng/mL
Time Frame: End of treatment
Population: Only patients who switched to one common dose, 300 mg od, are included in the AZD0837 analysis
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | AZD0837 | VKA, INR 2-3
Number analyzed (Participants) | 193 | 232
ng/mL | 68.9 [43.3 to 128.4] | 54.9 [31.9 to 99.0]

6. Secondary Outcome: Activated Partial Thromboplastin Time (APTT): Absolute Change From Baseline to End of Treatment
Description: Median Full range, Seconds
Time Frame: Baseline and End of treatment
Population: Only patients who switched to one common dose, 300 mg od, are included in the AZD0837 analysis
Measure: Median (Full Range); unit: sec
Arm/Group | AZD0837
Number analyzed (Participants) | 173
sec | 12.9 [-62 to 43]

7. Secondary Outcome: Electroconvulsive Therapy (ECT): Absolute Change From Baseline to End of Treatment
Time Frame: Baseline and End of Treatment
Population: Only patients who switched to one dose, 300 mg od, are included in the AZD0837 analysis
Measure: Median (Full Range); unit: sec
Arm/Group | AZD0837
Number analyzed (Participants) | 129
sec | 49.0 [-5 to 96]

8. Secondary Outcome: AZD0837: Plasma Concentration of AZD0837 at End of Treatment
Time Frame: End of treatment
Population: Only patients who switched to one dose, 300 mg od, are included in the AZD0837 analysis
Measure: Median (Full Range); unit: nmol/L
Arm/Group | AZD0837
Number analyzed (Participants) | 195
nmol/L | 675 [10 to 4090]

9. Secondary Outcome: AR-H067637XX, the Active Major Metabolite of AD0837: Plasma Concentration of AR-H067637XX, at End of Treatment
Time Frame: 154-711 days on treatment
Population: Only patients who switched to one dose, 300 mg od, are included in the AZD0837 analysis
Measure: Median (Full Range); unit: nmol/L
Arm/Group | AZD0837
Number analyzed (Participants) | 195
nmol/L | 341 [10 to 929]

ADVERSE EVENTS:
Time Frame: 154-711 days on treatment
Arm/Group | AZD0837 | VKA INR 2-3
Serious Adverse Events (participants affected / at risk) | 73/288 | 61/235
Other Adverse Events (participants affected / at risk) | 125/288 | 106/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD0837 (N=288) | VKA INR 2-3 (N=235)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 7 | 6
Atrial Fibrillation (Cardiac disorders) | 4 | 4
Angina Unstable (Cardiac disorders) | 0 | 3
Bradycardia (Cardiac disorders) | 3 | 2
Angina Pectoris (Cardiac disorders) | 2 | 1
Sick Sinus Syndrome (Cardiac disorders) | 2 | 1
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Atrial Flutter (Cardiac disorders) | 0 | 1
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Chordae Tendinae Rupture (Cardiac disorders) | 0 | 1
Coronary Artery Stenosis (Cardiac disorders) | 1 | 0
Heart Valve Incompetence (Cardiac disorders) | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 2
Eye Haemorrhage (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Retinal Artery Embolism (Eye disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 3
Gastric Ulcer (Gastrointestinal disorders) | 0 | 2
Abdominal Hernia (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1
Anal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Anal Ulcer (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Periodontal Disease (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 2 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 2
Asthenia (General disorders) | 1 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Jaundice Cholestatic (Hepatobiliary disorders) | 0 | 1
Corneal Graft Rejection (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 3
Erysipelas (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 3 | 3
Abscess Limb (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Intervertebral Discitis (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Foreign Body Trauma (Injury, poisoning and procedural complications) | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 2 | 1
Haemoglobin Decreased (Investigations) | 1 | 2
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 1
Blood Glucose Increased (Investigations) | 0 | 1
International Normalised Ratio Increased (Investigations) | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Inguinal Mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 0 | 2
Transient Ischaemic Attack (Nervous system disorders) | 1 | 2
Cerebral Artery Embolism (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1
Encephalitis (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Status Epilepticus (Nervous system disorders) | 1 | 0
Vascular Encephalopathy (Nervous system disorders) | 1 | 0
Vertebrobasilar Insufficiency (Nervous system disorders) | 1 | 0
Delusional Disorder, Persecutory Type (Psychiatric disorders) | 1 | 0
Dysthymic Disorder (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 0 | 1
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Arterial Occlusive Disease (Vascular disorders) | 1 | 0
Arterial Stenosis Limb (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0
Peripheral Artery Aneurysm (Vascular disorders) | 1 | 0
Peripheral Embolism (Vascular disorders) | 1 | 0
Subclavian Vein Thrombosis (Vascular disorders) | 1 | 0
800003Varicose Vein (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD0837 (N=288) | VKA INR 2-3 (N=235)
Diarrhoea (Gastrointestinal disorders) | 37 | 18
Flatulence (Gastrointestinal disorders) | 20 | 1
Oedema Peripheral (General disorders) | 25 | 20
Fatigue (General disorders) | 19 | 9
Nasopharyngitis (Infections and infestations) | 35 | 30
Bronchitis (Infections and infestations) | 14 | 18
Urinary Tract Infection (Infections and infestations) | 13 | 15
Fall (Injury, poisoning and procedural complications) | 4 | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 15 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 13
Dizziness (Nervous system disorders) | 24 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less